CLINICAL TRIAL: NCT06906835
Title: Efficacy of Reticulocyte Hemoglobin Equivalent-guided Versus Transferrin Saturation-guided Iron Supplement Protocol in Hemodialysis Patients: A Cluster Randomized Controlled Trial
Brief Title: Comparing Reticulocyte Hemoglobin and Transferrin Saturation to Guide Iron Treatment in People on Dialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Collaborators: Sysmex Asia Pacific (Industry); Center of Excellence for Metabolic Bone Disease in CKD patients, Faculty of Medicine, Chulalongkorn University (Unknown)
Responsible Party: Principal Investigator, Jeerath Phannajit, Chief, Division of Clinical Epidemiology, Department of Medicine, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0202/67
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hemodialysis; Anemia in End Stage Renal Disease
Keywords: Reticulocyte hemoglobin equivalent; Transferrin Saturation; Intravenous Iron Supplementation; Anemia in End Stage Renal Disease; Hemodialysis

STUDY DESIGN:
Intervention Model Description: Cluster randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RET-He-Guided Iron Supplementation (Experimental): Participants in this arm will receive intravenous (IV) iron therapy guided by reticulocyte hemoglobin equivalent (RET-He) levels.
  Interventions: Other: RET-He-Guided Iron Supplementation; Other: Common
- TSAT-Guided Iron Supplementation (Active Comparator): Participants in this arm will receive IV iron therapy guided by transferrin saturation (TSAT) and serum ferritin.
  Interventions: Other: TSAT-Guided Iron Supplementation; Other: Common

INTERVENTIONS:
Other: RET-He-Guided Iron Supplementation — Participants in this arm will receive intravenous (IV) iron therapy guided by reticulocyte hemoglobin equivalent (RET-He) levels.
  Iron dosing will follow a protocol based on RET-He values:
  * RET-He < 26 pg: IV iron 100 mg weekly
  * RET-He ≥ 26 pg and < 30 pg: IV iron 100 mg every 2 weeks
  * RET-He ≥ 30 pg and ≤ 36 pg: IV iron 100 mg every 4 weeks
  * RET-He > 36 pg or ferritin ≥ 800 ng/mL: Discontinue iron supplementation to prevent iron overload
  Arms: RET-He-Guided Iron Supplementation
Other: TSAT-Guided Iron Supplementation — Participants in this arm will receive IV iron therapy guided by transferrin saturation (TSAT) and serum ferritin, as per the Thai Clinical Practice Guidelines for Anemia in CKD (2021).
  Iron dosing will follow this TSAT-based protocol:
  * TSAT < 30% and ferritin < 200 ng/mL: IV iron 100 mg weekly
  * TSAT < 30% and ferritin 200-500 ng/mL: IV iron 100 mg every 2 weeks
  * TSAT < 30% and ferritin 500-800 ng/mL or TSAT 30-40%: IV iron 100 mg every 4 weeks
  * TSAT ≥ 40% or ferritin ≥ 800 ng/mL: Discontinue iron supplementation
  Arms: TSAT-Guided Iron Supplementation
Other: Common — All participants will receive erythropoiesis-stimulating agents (ESAs) according to a standardized dose adjustment protocol based on hemoglobin levels.
  Oral iron supplements will be discontinued.

SUMMARY:
The goal of this clinical trial is to find out which method is better for guiding iron treatment in adult patients with end-stage kidney disease (ESKD) on hemodialysis who have anemia.

The main questions it aims to answer are:

Can using reticulocyte hemoglobin equivalent (RET-He) to guide intravenous (IV) iron treatment be as effective as using transferrin saturation (TSAT)?

Does the method used to guide iron treatment affect outcomes such as death, heart problems, hospitalizations, infections, or the need for blood transfusions?

Researchers will compare RET-He-guided iron treatment with TSAT-guided iron treatment to see if RET-He works just as well and has similar or better outcomes.

Participants will:

Receive IV iron based on either RET-He or TSAT levels

Have blood tests done at the start, 3 months, and 6 months

Have their doses of iron and erythropoietin (a medication to treat anemia) adjusted based on the assigned protocol

Be monitored for clinical outcomes such as hospitalization, heart events, and infections

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18-80 years)
* ESKD on chronic hemodialysis ≥ 6 months
* EPO therapy ≥ 6 months
* Hb < 13.0 g/dL in male, < 12.0 g/dL in female

Exclusion Criteria:

* Serum ferritin > 800 ng/mL or TSAT > 40%
* Active infection or malignancy
* Hematologic disease including thalassemia major, hemolysis, myelofibrosis or myelodysplastic disease
* History of marrow suppressive or immunosuppressive medications in past 6 months
* History of active heart failure and recent myocardial infarction /stroke in past 6 months
* History of GI or external bleeding or receiving blood transfusion in past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Erythropoietin resistance index (ERI) [non-inferiority] | 6 months
  The erythropoietin resistance index (ERI, Unit/week/g/dL) is calculated by dividing the weekly body-weight-adjusted epoetin dose (international units per kilogram per week) by the hemoglobin concentration (grams per deciliter)
  The pre-specified non-inferiority margin is 20% (approx. 160 Unit/week/g/dL)
  Pre-specified subgroup analysis will be conducted: Patients with and without thalassemia trait will be separately analyzed

SECONDARY OUTCOMES:
All cause death | 6 months
Cardiovascular events | 6 months
  includes fatal and non-fatal acute coronary syndrome, stroke, and heart failure.
Blood Transfusions | 6 months
  Indication of blood transfusion will be decided by attending physicians for symptomatic anemia.
Hospitalizations | 6 months
  all non-elective admissions will be counted
Incidence of infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paweena Susantitaphong M.D, Ph.D., Study Chair — Center of Excellence for Metabolic Bone Disease in CKD patients, Chulalongkorn University; Jeerath Phannajit M.D., Study Director — Division of Clinical Epidemiology, Department of Medicine, King Chulalongkorn Memorial Hospital, Thai Red Cross; Chalermchon Suttaluang M.D., Principal Investigator — Division of Nephrology, Department of Medicine, King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathumwan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD are planned to be shared with a reasonable and relevant reason, please contact investigator.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Chinudomwong P, Binyasing A, Trongsakul R, Paisooksantivatana K. Diagnostic performance of reticulocyte hemoglobin equivalent in assessing the iron status. J Clin Lab Anal. 2020 Jun;34(6):e23225. doi: 10.1002/jcla.23225. Epub 2020 Feb 11. PMID 32043622
- [Background] Susantitaphong P, Siribumrungwong M, Takkavatakarn K, Chongthanakorn K, Lieusuwan S, Katavetin P, Tiranathanagul K, Lekhyananda S, Tungsanga K, Vanichakarn S, Eiam-Ong S, Praditpornsilpa K. Effect of Maintenance Intravenous Iron Treatment on Erythropoietin Dose in Chronic Hemodialysis Patients: A Multicenter Randomized Controlled Trial. Can J Kidney Health Dis. 2020 Jun 19;7:2054358120933397. doi: 10.1177/2054358120933397. eCollection 2020. PMID 32612843
- [Background] Babitt JL, Eisenga MF, Haase VH, Kshirsagar AV, Levin A, Locatelli F, Malyszko J, Swinkels DW, Tarng DC, Cheung M, Jadoul M, Winkelmayer WC, Drueke TB; Conference Participants. Controversies in optimal anemia management: conclusions from a Kidney Disease: Improving Global Outcomes (KDIGO) Conference. Kidney Int. 2021 Jun;99(6):1280-1295. doi: 10.1016/j.kint.2021.03.020. Epub 2021 Apr 8. PMID 33839163
- [Background] Wish JB, Anker SD, Butler J, Cases A, Stack AG, Macdougall IC. Iron Deficiency in CKD Without Concomitant Anemia. Kidney Int Rep. 2021 Aug 10;6(11):2752-2762. doi: 10.1016/j.ekir.2021.07.032. eCollection 2021 Nov. PMID 34805628